CLINICAL TRIAL: NCT01745705
Title: Immediate Effects of Cervical Spine Manipulation on Balance and Joint Proprioception in Healthy Individuals
Brief Title: Cervical Spine Manipulation Affects on Balance and Proprioception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Emilio, Assistant Professor, University of Nevada, Las Vegas
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1105-3780
Record Dates: First submitted 2012-12-05; First posted 2012-12-10 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Neck Pain; Headache
Keywords: Manipulation; Balance; Proprioception
MeSH Terms: conditions — Neck Pain; Headache

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cervical Spine Manipulation (Experimental): Subjects will lie supine on a treatment table and receive a high velocity low amplitude thrust joint manipulation to their cervical spine in rotation to each side of the neck.
  Interventions: Other: Cervical Spine Manipulation
- Manual Contact (Sham Comparator): Subjects will lie supine on a treatment table and have their suboccipital region gently cupped by the therapist for 30 seconds. No movement or force will be applied, just simple manual contact.
  Interventions: Other: Manual Contact

INTERVENTIONS:
Other: Cervical Spine Manipulation
  Arms: Cervical Spine Manipulation
Other: Manual Contact
  Arms: Manual Contact

SUMMARY:
Cervical spine manipulation (CSM) is utilized by many health care practitioners in the management of patients with neck pain and headache. How CSM works is not understood however, most researchers agree that there is likely a combination of mechanical, neurophysiological and placebo effects. This study will test for possible neurophysiological effects by examining for changes in a person's ability to reposition their head and neck in space, and maintain their balance following CSM.

DETAILED DESCRIPTION:
Consenting participants will have their proprioception tested through a joint repositioning error test for their cervical spine, and also have their balance tested through a Neurocom Balancemaster. Following these pre-intervention measures, they will receive in a random order, either a cervical spine manipulation (CSM) or a sham manipulation, and then have tests repeated to analyze for changes and differences between interventions.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals between the ages of 18 and 60

Exclusion Criteria:

* current neck pain/symptoms; neck pain symptoms within the last 6 months; confirmation or possibility of pregnancy; dizziness; vertigo, or nausea; history of cervical spine surgery; rheumatoid arthritis; osteoporosis; osteopenia; ankylosing spondylitis; cancer; or vertebral artery insufficiency.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2011-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Cervical joint proprioception | 1 day (Immediately after the intervention)
  Subjects wear a headband with a mounted laser pointer and sit 1 meter away from a wall. They assume their comfortable neutral cervical posture and then close their eyes and extend their cervical spine and return to their neutral posture with eyes closed. The laser pointer marks the point of return and we measure the difference between start and end points for error.

OTHER OUTCOMES:
SMART Neurocom Balance Master | 1 day (Immediately after the intervention)
  Subjects stand on a force plate on a SMART Neurocom Balance Master and complete a Sensory Organization Test (SOT) program which assesses somatosensory, visual and vestobular systems used in maintaining balance.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy, University of Nevada Las Vegas, Las Vegas, Nevada, United States

REFERENCES:
- See also: Related Info — http://pt.unlv.edu/louie.htm